CLINICAL TRIAL: NCT01954563
Title: A Phase I Trial Evaluating Mucosal Administration of a Candidate TB Vaccine, MVA85A, as a Way to Induce Potent Local Cellular Immune Responses and Avoid Anti-vector Immunity
Brief Title: Study Evaluating Aerosol and Intradermal Administration of a Candidate Tuberculosis (TB) Vaccine, MVA85A, as a Way to Increase Immune Response and Avoid Anti-vector Immunity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB035
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine; Immunogenicity
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Receive 5x10^7 MVA85A by aerosol at day 0, followed by boost intradermal vaccination of 5x10^7 MVA85A at day 28.
  Interventions: Biological: MVA85A
- Group 2 (Experimental): Receive 5x10^7 MVA85A by intradermal injection at day 0, followed by boost aerosol vaccination of 5x10^7 MVA85A at day 28.
  Interventions: Biological: MVA85A
- Group 3 (Experimental): Receive 5x10^7 MVA85A by intradermal injection at day 0, followed by boost intradermal vaccination of 5x10^7 MVA85A at day 28.
  Interventions: Biological: MVA85A

INTERVENTIONS:
Biological: MVA85A — Modified vaccinia virus Ankara (MVA) is a highly attenuated strain of vaccinia with an antigen 85A insert.

SUMMARY:
Boost vaccinations sometimes have no effect because the body has got used to the vaccine and no longer reacts to it. We are therefore investigating whether vaccinating with aerosolised MVA85A (a candidate tuberculosis vaccine) followed by a boost MVA85A intradermal vaccination (or vice versa) avoids this and increases the immune response to vaccination.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to enter the trial:

* Healthy adult aged 18-55 years
* Resident in or near Oxford for the duration of the trial period
* No relevant findings in medical history or on physical examination
* Confirmation of prior vaccination with BCG not less than 6 months prior to projected trial vaccination date (by visible BCG scar on examination or written documentation)
* Allow the Investigators to discuss the individual's medical history with their GP
* Use effective contraception for the duration of the trial period (females only)
* Refrain from blood donation during the trial
* Give written informed consent
* Allow the Investigator to register subject details with a confidential database to prevent concurrent entry into clinical trials
* Able and willing (in the Investigator's opinion) to comply with all the trial requirements

Exclusion Criteria:

Subjects must meet none of the following criteria to enter the trial:

* Any respiratory disease, including asthma
* Current smoker
* Clinically significant abnormality on screening chest x-ray
* Clinically significant abnormality of pulmonary function tests
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy
* Current use of any medication taken through the nasal or inhaled route including cocaine or other recreational drugs
* Laboratory evidence at screening of latent M. tb infection as indicated by a positive ELISPOT response to ESAT6 or CFP10 antigens
* Clinical, radiological, or laboratory evidence of current active TB disease
* Previous vaccination with candidate vaccine MVA85A or candidate vaccine FP85A or any other recombinant MVA vaccine
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* History of serious psychiatric condition
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine, sedative drugs, or any local or general anaesthetic agents
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the subject in the trial
* Positive HBsAg, HCV or HIV antibodies
* Female currently lactating, confirmed pregnancy or intention to become pregnant during trial period
* Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device other than the trial vaccine for 30 days prior to dosing with the trial vaccine, or planned use during the trial period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the subject at risk or may influence the result of the trial or may affect the subject's ability to participate in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety of 5 x 10^7 pfu dose of MVA85A administered by aerosol and compared to the same dose administered intradermally | 24 weeks from enrolment
  Actively and passively collected data on adverse events

SECONDARY OUTCOMES:
Immunogenicity of 5 x 10^7 pfu dose of MVA85A administered by aerosol followed by the same dose administered intradermally, compared to the same dose of MVA85A given intradermally and boosted by aerosol | 24 weeks from enrolment
  * Characterise mucosal and systemic immunogenicity of viral vector (MVA) and insert (Ag85A) by comprehensive characterisation of humoral and cellular immune responses
  * Evaluate functional relevance of anti-vector immunity induced by aerosol and systemic immunisation in MVA85A-prime followed by homologous MVA85A-boost administered 4 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Manjaly Thomas ZR, Satti I, Marshall JL, Harris SA, Lopez Ramon R, Hamidi A, Minhinnick A, Riste M, Stockdale L, Lawrie AM, Vermaak S, Wilkie M, Bettinson H, McShane H. Alternate aerosol and systemic immunisation with a recombinant viral vector for tuberculosis, MVA85A: A phase I randomised controlled trial. PLoS Med. 2019 Apr 30;16(4):e1002790. doi: 10.1371/journal.pmed.1002790. eCollection 2019 Apr. PMID 31039172
- See also: Jenner Institute Clinical Trials — http://www.jenner.ac.uk/clinicaltrials